CLINICAL TRIAL: NCT04909658
Title: The Effect of Acceptance and Commitment Therapy for Improving Psychological Well-being in Parents of Individuals With Autism Spectrum Disorder: a Randomized Controlled Trial
Brief Title: The Effect of Acceptance and Commitment Therapy
Acronym: ASDMatrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.Anna Rehabilitation Institute (Other)
Collaborators: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CNR-AMMCEN 54444/2018
Record Dates: First submitted 2021-04-22; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Autism, Infantile
Keywords: Autism spectrum disorder; Psychological well-being
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Psychological Well-Being | interventions — CAMFTP protocol

STUDY DESIGN:
Intervention Model Description: A single-blind, randomized controlled study was conducted at our CNR center in Messina. The first stage was based on the recruitment of the parents for the study. Next, the eligible individuals underwent a clinical examination at baseline [T0]. In the third stage, participants were randomly assigned to two groups using a computer-generated randomization code. The following people were all blinded to the group membership of the parents: the physicians (who carried out the clinical baseline assessment [T0] and post-treatment investigation [T1]), the primary researchers, and the data entry assistants. In the fourth stage, participants underwent ACT or PT training therapies. Treatments were carried on by expert therapists who were blinded to all clinical information and also to the aim of the study. At the end of treatment, participants from both groups were given a final evaluation [T1], using the same protocol as at a baseline.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The following people were all blinded to the group membership of the parents: the physicians (who carried out the clinical baseline assessment [T0] and post-treatment investigation [T1]), the primary researchers, and the data entry assistants. In the fourth stage, participants underwent ACT or PT training therapies. Treatments were carried on by expert therapists who were blinded to all clinical information and also to the aim of the study. At the end of treatment, participants from both groups were given a final evaluation [T1], using the same protocol as at a baseline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT matrix protocol (Experimental): Parents of childrens with Autism Spectrum Disorders (ASD). The ACT protocol group received exercises to improve the psychological well-being of the parents.
  Interventions: Behavioral: ACT Matrix
- PT protocol (Active Comparator): Parents of childrens with Autism Spectrum Disorders (ASD).
  Interventions: Behavioral: PT Protocol

INTERVENTIONS:
Behavioral: ACT Matrix — The ACT protocol group performs exercises to improve the psychological well-being of parents. The matrix is an ACT protocol that is usually presented visually to patients and consists of two intersecting lines that make up four quadrants, which provide a "point of view" on one's psychological actions and experiences. The vertical line is the line of experience, the upper part corresponds to the experience of life linked to the five senses - sight, hearing, taste, smell and touch - (experience of the five senses), the lower part refers to the experiences internal as thoughts and feelings (internal/mental experience). The horizontal line is the behavior line, the left side concerns the actions that perform the function of moving us away from experiences, emotions, unwanted thoughts (experiential avoid-ance), the right side indicates the actions we take to get closer and go towards our values (committed action).
  Arms: ACT matrix protocol
Behavioral: PT Protocol — The PT protocol group received behavioral tasks related to child management. Parent training interventions carried out in groups can be a good solution to modify parent behavior by providing social support and new coping strategies. The intervention includes 24 weekly meetings lasting 90 minutes each. The total intervention is six months.
  Arms: PT protocol

SUMMARY:
In this randomized control study, investigators will evaluate the effectiveness of the Acceptance and Commitment Therapy (ACT) matrix behavioral protocol compared to Parent Training (PT) programs in improving the psychological well-being of parents of children with Autism Spectrum Disorder (ASD). Twelve parents will be randomly and equitably assigned to two matched groups in which individuals will undergo 24 weekly ACT (experimental group) or conventional PT (control group) protocol meetings

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a lifelong neurodevelopmental disorder characterized by core deficits in maladaptive behaviors, communication skills, and self-regulation im-pairments affecting the socio-relational performance of children, but also of their parents. It has widely been demonstrated that raising a child with autism involves chronic challenges consistently associated with high levels of psychological distress. Often parents become isolated from family and friends who may not understand the child's be-havior and disability. The chronic stress experienced by parents of children with ASD also reported to be greater than those experienced by parents of children with other disabilities, such as Down Syndrome, behavioral disorders and Fragile X Syndrome, and also associated with increased divorce rates.

It is clear that family members, in this condition, should be supported in the development of new parenting skills useful to achieve targets of intervention while reducing psycho-logical distress. Indeed, reinforcement of parental resources has been considered as potential mediating factors of ASD treatment, which may reduce maladaptive behaviors in children. The present single-blind Randomized Controlled Trial (RCT) is aimed to compare, for the first time, the efficacy of the ACT approach in ASD parents with respect to the PT. Several papers reported the beneficial effects of PT groups as classic support to increase parenting skills in managing the behavior of children with ASD while reducing parental stress. Nevertheless, none has evalu-ated if ACT may be a more powerful approach to threat psychological reaction to the stress of caring for ASD children. The investigators hypothesized that psychological difficulties of parents of children with autism could decrease after a course with goals of transmitting behavioral educational techniques and promoting psychological adjustment through defusion and acceptance strategies. Primary outcome measures and secondary outcome measures will be collected. A pre/post-treatment assessment will be conducted regarding the measurement and change in parental psychological flexibility during the intervention. The primary outcome measures that will be used are the Acceptance and Action Questionnaire II (AAQ-II) to measure the person's psychological flexibility and ability to stay in touch with emotions and the Home Situation Questionnaire (HSQ-ASD) which give objective measures of the perception and influence of children's behavior in the parents' lives. Secondary outcome measures will be the Valued Living Questionnaire (VLQ) to identify areas important to the person, the Mindfulness Attention Awareness Scale (MAAS) which measures an individual's tendency toward intentional awareness, and the Parental Stress Index (PSI) to assess pre- and post-treatment stress levels.

ELIGIBILITY:
The families were recruited as part of an ongoing research program and tested at our clinical facilities.

Inclusion criteria were based on children characteristics as follows:

* between 3 and 13 years of age;
* clinical diagnosis of ASD based on the DSM-5 criteria from a licensed clinical child neuropsychiatrist;
* DSM-5 severity scores from mild (level 1) to moderate (level 2) in both social communication and restricted interests and repetitive behaviors domains;
* a verbal and performance Developmental Quotient: Griffiths Mental Development Scales, Extended Revised: 2 to 8 years (GMDS-ER 2-8 Luiz et al. 2006) and Wechsler Intelligence Scale for Children (WISC-IV Wechsler D. 2003) above 70;
* no hearing, visual, or physical disabilities that would prevent participation in the intervention;
* not being on psychiatric medication. All children have a previous diagnosis that was further confirmed through the assessment and the consensus of experienced professionals on the research team (i.e., a child neuropsychiatrist and a clinical psychologist).

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Acceptance and Action Questionnaire (AAQ-II) | 6 months after the admission assessment
  The AAQ-II is a ten-item test with answers on a scale from 1 (never true) to 7 (always true) to measure the person's psychological flexibility and their ability to stay in touch with emotions. The items focus on the willingness to separate unwanted private events, on the ability to live in the present moment and on the commitment to adopt flexible and valuable actions during the experience of internal negative events.
Home Situation Questionnaire (HSQ-ASD) | 6 months after the admission assessment
  The HSQ-ASD is a caregiver-rated scale designed to assess the severity of disruptive and non-compliant behaviors in children. The score obtained with this scale refers to the parent's perception of their child's behavioral manifestations. Within the scale, data are collected on inflexibility and avoidance manifested by the child. This modified and revised version for ASD consists of 27 elements. Parents are asked to indicate if their children have problems with compliance in these situations and, if so, to rate severity on a Likert scale of 0 to 9, with higher scores indicating greater non-compliance.

SECONDARY OUTCOMES:
Valued Living Questionnaire (VLQ) | 6 months after the end of treatment
  The VLQ is a questionnaire exploring some areas of life that people consider important such as family relationships; marriage/couple; intimate relationships; friends; social relationships; work; culture/training; leisure/entertainment; spirituality; civic commitment/community life and self-care.
  The questionnaire provides an importance score, in which, for each dimension, the person is asked to rate on a scale from 1 (not at all important) to 10 (extremely important) how important that area of their life is.
Mindful Attention Awareness Scale (MAAS) | 6 months after the end of treatment
  The Mindful Attention Awareness Scale [MAAS] measures individual differences in daily awareness states. Then, respondents rated the 15 elements of the scale on a 7-point Likert-type scale, from 1 (almost always) to 7 (almost never). Higher values indicate higher levels of awareness.
Parental Stress Index/Short Form (PSI/SF) | 6 months after the end of treatment
  The PSI/SF is a self-assessment questionnaire. The administration and compilation of the test take about 10-15 minutes. The hypothesis underlying the test is that parental stress levels are given by the interaction of 3 different factors: 1 characteristic of the children, 2 characteristics of the parent, 3 aspects related to the parental situation.The short form is composed of 36 items, divided into three subscales: (1) Parental Distress (PD), which taps into parental feelings; (2) Parent-Child Dysfunctional Interaction (P-CDI), which focuses on the perception of the child as not responding to parental ex-pectations; (3) Difficult Child (DC), which is centered on some of the characteristics of the child that make it easy or difficult to manage.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB), Messina, Italy

REFERENCES:
- [Background] Bearss K, Johnson C, Smith T, Lecavalier L, Swiezy N, Aman M, McAdam DB, Butter E, Stillitano C, Minshawi N, Sukhodolsky DG, Mruzek DW, Turner K, Neal T, Hallett V, Mulick JA, Green B, Handen B, Deng Y, Dziura J, Scahill L. Effect of parent training vs parent education on behavioral problems in children with autism spectrum disorder: a randomized clinical trial. JAMA. 2015 Apr 21;313(15):1524-33. doi: 10.1001/jama.2015.3150. PMID 25898050
- [Background] Bond FW, Bunce D. Mediators of change in emotion-focused and problem-focused worksite stress management interventions. J Occup Health Psychol. 2000 Jan;5(1):156-63. doi: 10.1037//1076-8998.5.1.156. PMID 10658893
- [Result] Abbeduto L, Seltzer MM, Shattuck P, Krauss MW, Orsmond G, Murphy MM. Psychological well-being and coping in mothers of youths with autism, Down syndrome, or fragile X syndrome. Am J Ment Retard. 2004 May;109(3):237-54. doi: 10.1352/0895-8017(2004)1092.0.CO;2. PMID 15072518